CLINICAL TRIAL: NCT07080775
Title: A Phase I Clinical Study on the Safety and Tolerability of iPSC-Derived Dopaminergic Neural Progenitor Cell Injection Via Stereotaxic Brain Transplantation for the Treatment of Primary Parkinson's Disease
Brief Title: The Safety and Tolerability of XS411CN Injection in Treatment of Primary Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: XellSmart Bio-Pharmaceutical (Suzhou) Co., Ltd. (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XS411-Allo-LOPD-CN1/2-P01
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4.5×10^6 cells / bilateral putamen (Experimental)
  Interventions: Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection
- 9.0×10^6 cells / bilateral putamen (Experimental)
  Interventions: Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection
- 1.8×10^7 cells / bilateral putamen (Experimental)
  Interventions: Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection

INTERVENTIONS:
Drug: human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection — 5.0×10^7 cells/mL, injection, once, 12 months

SUMMARY:
This Phase I clinical trial is designed to evaluate the safety, tolerability of a single dose of XS411 (derived dopaminergic neural progenitor cell injection) in patients with primary Parkinson's disease

DETAILED DESCRIPTION:
This is a phase I clinical study to evaluate the safety and tolerability of human allogeneic induced pluripotent stem cell (iPSC)-derived dopaminergic neural progenitor cell injection (XS411CN) via brain stereotactic transplantation for the treatment of primary Parkinson's disease.

The study adopts a single-arm, open-label, non-randomized dose-escalation design to evaluate the safety, tolerability, and preliminary efficacy of stereotactic brain transplantation of XS411CN in patients with primary Parkinson's disease and explore the optimal recommended dose. 12 to 18 patients with primary Parkinson's disease are planned to be enrolled.

On the day of cell transplantation surgery, the planned dose of XS411CN is transplanted into the bilateral putamen of the subjects by brain stereotactic technology.

After receiving the XS411CN transplantation, the subjects will receive immunosuppressants. All subjects receive standard treatment at the same time.

Each patient receives a safety observation period of 28 days after cell transplantation with XS411CN. This study adopts the traditional "3+3 " dose escalation method. The trial starts with a low dose and the dose will be increased gradually. Each subject will be closely observed for 7 days after surgery, and the dose-limiting toxicity (DLT) events that may occur within 28 days after the first transplant treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 50 and 75 years old;
2. Diagnosed as 'clinically established PD' consistent with MDS clinical Diagnostic Criteria for Parkinson's disease,
3. A minimum of 5 years since diagnosis;
4. Hoehn- Yahr score during the off-time is 3 to 4;
5. The subjects with an average of at least 2.5 hours of "off time" per day;
6. Stable anti-PD therapy for at least 1 month before screening;
7. Anti-PD treatment was once effective, but the efficacy has declined significantly or drug-induced motor complications have occurred, affecting the quality of life;
8. Positive levodopa challenge test (MDS-UPDRS-III score improvement from off- state to on- state > 30%);
9. At least three months before the first administration, the subject should have completed all vaccinations as recommended by local authorities;
10. The results of complete blood count meet the following conditions: ANC ≥ 2.0×109 /L, WBC ≥ 4.0×109 /L, PLT≥ 100×109 /L, HGB ≥ 10g/dL
11. The patient or his/her legal guardian agree to accept the study and signed the informed consent form in writing.

Exclusion Criteria:

1. Parkinsonian syndrome or secondary Parkinson's disease (Atypical Parkinson's syndrome (Parkinson's plus syndrome, secondary Parkinson's syndrome, hereditary degenerative Parkinson's syndrome);
2. Patients are in advanced stages of Parkinson's disease and are experiencing severe, disabling peak-dose dyskinesia or biphasic dyskinesia and/or unpredictable or widely fluctuating symptoms;
3. Severe cognitive impairment (MMSE<24, poor compliance due to dementia, inability to accurately record diaries, and/or inability to sign informed consent;
4. Those with a history of severe mental illness, or those with severe suicidal tendencies as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS), or those with suicidal ideation in the past 12 months, or those who have attempted suicide in the past 5 years;
5. Patients with severe brain atrophy, space-occupying lesions, hydrocephalus, cerebral vascular malformations as indicated by head CT/MRI, and those with structural abnormalities that may affect transplantation or increase surgical risks as determined by the investigators;
6. Currently with active internal bleeding; or arterial puncture at a site that is difficult to stop bleeding within 1 week before screening; or gastrointestinal or urinary bleeding within 3 weeks before screening;
7. History of striatal or extrapyramidal surgery, including but not limited to deep brain stimulation (DBS) surgery and globus pallidus lesion;
8. Coagulation abnormalities;
9. Abnormal liver and kidney function laboratory tests during the screening period;
10. The patient is currently receiving or has previously received the following treatments:

    * Use of benzodiazepines at a dose level equal to or higher than the recommended dose in Package Insert for more than 4 weeks cumulatively since one month before enrollment, immunosuppressants (except for the immunosuppressants to be used in this study), or antipsychotics within 3 months before treatment;
    * Use of botulinum toxin, phenol, subarachnoid baclofen injection, or interventional treatment for dystonia or spasticity within 6 months before treatment;
    * Have a history of epilepsy or use anti-epileptic drugs for prevention;
    * Received cell therapy within 3 months before screening;
11. Contraindications to general anesthesia or stereotactic surgery (such as sleep apnea, chronic obstructive pulmonary disease, etc.), MRI or PET examinations;
12. Those with the following abnormalities in the past or detected (if any of the following is met, they will be excluded):

    * Evidence of congestive heart failure or history of end-stage cardiovascular disease;
    * Severe arrhythmias and poorly controlled arrhythmias;
    * Clinically significant electrocardiogram abnormalities during the screening or baseline period;
    * History of unstable angina or acute myocardial infarction within the past 3 months;
    * Diabetic patients with poor glycemic control;
    * Hypertensive patients with poorly controlled blood pressure;
13. Patients with active infection during the screening period (except mild local skin infection) that need antibiotic, antifungal, or antiviral treatment but infection is still not under control;
14. The presence of severe lung diseases during the screening period;
15. Patients with uncontrolled autoimmune diseases;
16. During the screening period, patients have severe arthritis, limp, severe sequelae of stroke, severe osteoporosis, or history of severe trauma within 1 month, etc., which the investigators assess may affect the evaluations;
17. Any history of malignancy, excluding cured basal cell carcinoma and/or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or ductal carcinoma of the breast;
18. Serious infectious diseases;
19. Pregnant or lactating women, women who plan to become pregnant during the study and within 6 months after the end of the study, or women who are unwilling to use effective contraceptive measures;
20. Patients who have participated in other clinical studies of drugs or medical devices within 3 months before treatment;
21. Have a long history of alcoholism or drug abuse;
22. Patients with a history of severe allergies or allergies to investigational drugs and immunosuppressants;
23. Any other conditions that the investigator considers unsuitable for participation in the study.
24. Severe depression
25. Hallucinations, and hallucinations still exist after optimizing Parkinson's medications
26. Patients have undergone MRI-guided focused ultrasound thalamotomy
27. Used immunosuppressants within 3 months, except for the immunosuppressants to be used in this study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of XS411CN in treatment of primary Parkinson's disease | 28 days after administration of XS411CN
  To evaluate the safety and tolerability of XS411CN in treatment of primary Parkinson's disease through:
  1）The occurrence and incidence of adverse events and serious adverse events (adverse event grading criteria are based on NCI-CTCAE V5.0) 28 days after administration of XS411CN; 2) Changes in vital signs, laboratory tests, 12-lead electrocardiogram, etc. compared with baseline after administration of XS411CN;

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes